CLINICAL TRIAL: NCT03732664
Title: ICIs Neoadjuvant Therapy in Resectable Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2018-10-29; First posted 2018-11-06 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2021-10

CONDITIONS: High-Risk Resectable NSCLC
MeSH Terms: interventions — Nivolumab; pembrolizumab; toripalimab; sintilimab; tislelizumab; durvalumab

STUDY DESIGN:
Intervention Model Description: Anti-PD-1 or anti-PD-L1 antibody administration:
  One to four doses of anti-PD-1 or anti-PD-L1 antibody will be administered to enrolled patients on Day -56, Day -42, Day -28, and Day-14 (+/- two days) prior to planned surgery on Day 0 or up to +10 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Drug: Nivolumab, Pembrolizumab, Toripalimab, Sintilimab, Sintilimab, Tislelizumab, Durvalumab

INTERVENTIONS:
Drug: Nivolumab, Pembrolizumab, Toripalimab, Sintilimab, Sintilimab, Tislelizumab, Durvalumab — One to four doses of anti-PD-1 or anti-PD-L1 antibody will be administered to enrolled patients on Day -56, Day -42, Day -28, and Day-14 (+/- two days) prior to planned surgery on Day 0 or up to +10 days.
  Other Names: BMS-936558; MDX1106; Keytruda

SUMMARY:
The proposed study will evaluate the safety and feasibility of preoperative administration nivolumab in patients with high-risk resectable NSCLC, and will facilitate a comprehensive exploratory characterization of the tumor immune milieu and circulating immune cells and soluble factors in these patients. Data obtained in this study will provide valuable information for planning further prospective clinical trials of anti-PD-1 or anti-PD-L1 in NSCLC, both in the peri-operative and advanced disease setting.

DETAILED DESCRIPTION:
The proposed study will evaluate the safety and feasibility of preoperative administration nivolumab in patients with high-risk resectable NSCLC, and will facilitate a comprehensive exploratory characterization of the tumor immune milieu and circulating immune cells and soluble factors in these patients. Data obtained in this study will provide valuable information for planning further prospective clinical trials of anti-PD-1 or anti-PD-L1 in NSCLC, both in the peri-operative and advanced disease setting. Ultimately, it is highly desirable to discover prospective biomarkers of response and toxicity to allow patients with NSCLC who are most likely to derive benefit to receive anti-PD-1 or anti-PD-L1 treatment, and conversely to minimize the risk of toxicity and ineffective treatment for patients who are unlikely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small-cell lung cancer (core biopsy required).

  * Squamous or non-squamous histology.
  * Diagnostic core biopsy specimens must be reviewed by a faculty pathologist at The Second Affiliated Hospital Zhejiang University School of Medicine.
  * Either a formalin fixed paraffin block or a minimum of fifteen 5-micron tissue sections (slides) of tumor biopsy sample must be available for biomarker evaluation (study pathologist must review for adequacy of sampling). This can be obtained from archived tissues, or from a new biopsy if needed.
* Stage - High risk NSCLC with resection option for potential cure, as assessed by a faculty surgeon at The Second Affiliated Hospital Zhejiang University School of Medicine. This may include clinical stage IA3 (≥2cm), II and IIIA(see Appendix A). Subjects with N3 nodal involvement are not included.
* ECOG performance status 0-1.
* Adequate organ function as follows:

  * Leukocytes ≥ 2,000/mm3.
  * Absolute neutrophil count (ANC) ≥ 1000/mm3.
  * Platelet count ≥ 100,000/mm3.
  * Hemoglobin ≥ 9 g/dL.
  * Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL.

Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL.

* Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
* AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 3 times the upper limit of normal.

  * Subjects must have adequate lung function to permit surgical resection determined by pre-enrollment pulmonary function tests to include DLCO.
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for up to 23 weeks after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for up to 31 weeks after the last dose of nivolumab. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of registration. Women must not be breastfeeding.
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines must be obtained before the performance of any protocol related procedures that are not part of normal patient care. Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs.

Exclusion Criteria:

* Subjects are excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Subjects are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. As there is potential for hepatic toxicity with nivolumab or nivolumab/ipilimumab combinations, drugs with a predisposition to hepatoxicity should be used with caution in patients treated with nivolumab-containing regimen.
* Administration of chemotherapy or any other cancer therapy in the pre-operative period.
* Subjects with active concurrent malignancies are excluded i.e. cancers other than NSCLC (except non melanoma skin cancers, in situ bladder, gastric, breast, colon or cervical cancers/dysplasia).
* Subjects with brain metastasis are excluded from this study, and all patients should have brain imaging (either MRI brain or CT brain with contrast) prior to enrollment.
* Subjects with a history of symptomatic interstitial lung disease.
* Active systemic infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* Known positive history or positive test for Human Immunodeficiency Virus or
* Acquired ImmunoDeficiency Syndrome (AIDS).
* History of allergy to study drug components.
* Women who are pregnant or nursing.
* Men with female partners (WOCBP) that are not willing to use contraception.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-regulatory pathways).
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Safety and Adverse effects | 8 weeks
  Safety will be measured by drawing safety labs. (CBC and a Chemistry Panel will be drawn at 2 week intervals during Nivolumab administration). Grade 3 and 4 lab abnormalities will be recorded from both participating sites. Safety will also be measured by recording Grade 3 and 4 CTCAE 4.03 listed adverse events that occur while a subject is participating in the study.

SECONDARY OUTCOMES:
Rate of Enrollment | 8 weeks
  Feasibility will be measured by the rate of enrollment of the 40 subjects at the 2 sites.
Pathologic Response | 6 weeks
  To assess pathologic response to neoadjuvant nivolumab in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy.
Radiographic Response | 5 weeks
  To assess radiographic response to neoadjuvant nivolumab using RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Derived] Chen Y, Shao Z, Hao Z, Xin Z, Chen X, Huang L, Chen D, Lin M, Liu Q, Xu X, Li J, Wu D, Yan J, Chai Y, Wu P. Epithelium/imcDC2 axis facilitates the resistance of neoadjuvant anti-PD-1 in human NSCLC. J Immunother Cancer. 2024 Aug 12;12(8):e007854. doi: 10.1136/jitc-2023-007854. PMID 39134346